CLINICAL TRIAL: NCT06756737
Title: The Application of 68Ga-Pentixafor Alongside 68Ga-FAPI-04 PET/MR for Assessing Primary Aldosteronism.
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHE-2024089
Record Dates: First submitted 2024-11-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Primary Aldosteronism
Keywords: PET/CMR; Primary aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Research group: This study aims to recruit 30 patients with primary aldosteronism.
- Control group: The study included 30 patients with primary hypertension as the control group.

SUMMARY:
The objective of this observational study is to utilize the advantages of 68Ga-Pentixafor subtyping diagnosis and the diagnostic ability of 68Ga-FAPI-04 for cardiovascular disease to identify primary aldosterone patients in need of adrenal surgery using non-invasive methods, while also assessing the degree of myocardial injury. Providing new, simple, and comprehensive diagnostic approaches for patients with primary aldosteronism, and improving the accuracy of clinical decision-making, can help develop personalized treatment plans in the early stages, thereby improving the long-term prognosis of primary aldosteronism patients.

DETAILED DESCRIPTION:
Hypertension, as a global clinical problem, seriously endangers public health. According to the latest report from the World Health Organization, approximately 1.28 billion adults aged 30 to 79 worldwide suffer from hypertension, mainly concentrated in low- and middle-income countries. According to the latest data released by the National Cardiovascular Disease Center of China, the prevalence of hypertension among adults aged 18 and above in China is as high as 27.5%, with a staggering 245 million patients, and the patient population is becoming younger. For a long time, hypertension has been regarded as the second leading risk factor for increasing global mortality rates, imposing a heavy burden on society and the economy. It is estimated that hypertension causes economic losses of over 200 billion yuan annually in China. In this context, primary aldosteronism (PA) has attracted much attention as a high-risk and treatable hypertension disease. Aldehydes are caused by adrenal cortex lesions, accounting for 5% -12% of newly diagnosed hypertension patients, and up to 20% of refractory hypertension patients. It is estimated that there are at least 12 million aldehyde patients in China. The mortality rate of aldehyde patients is higher than that of primary hypertension patients matched for age, gender, and blood pressure. Timely diagnosis and targeted treatment of patients with aldosterone can not only help alleviate or cure hypertension, but also reduce the damage of aldosterone itself to target organs such as the heart and kidneys, lower the incidence of complications, significantly improve patient's quality of life, and ultimately reduce mortality rates. Therefore, studying the diagnosis and treatment of aldehydes is not only necessary for medical research, but also a significant contribution to public health. PA is a complex disease with multiple subtypes and etiologies. In theory, surgical removal of adrenal cortex lesions can effectively control or even cure hypertension. However, in practice, the effectiveness of surgical treatment for some patients is not ideal, especially with poor long-term prognosis and a high risk of blood pressure relapse. Not all PAs have the potential for surgical treatment. As recommended by the guideline from the Journal of the American College of Cardiology, Aldehyde can be divided into two categories based on treatment: surgical cure and surgical non-cure. Laparoscopic unilateral adrenalectomy is the preferred treatment method for the surgical curable group, while non-surgical patients are usually treated with drugs such as mineralocorticoid receptor antagonists. Compared with patients who undergo surgical treatment, those who receive medication have a higher incidence of atrial fibrillation, so it is important to detect as many patients as possible who are suitable for surgical treatment. Therefore, accurate classification diagnosis is crucial for selecting treatment methods and achieving personalized treatment. The bottleneck in improving the cure rate of hypertension after adrenal surgery in patients with primary aldosteronism lies in the many limitations of current classification diagnostic tools. The conventional classification and diagnostic methods for aldehyde include anatomical imaging such as Computed Tomography(CT) or Magnetic Resonance Imaging(MRI) and adrenal vein sampling (AVS), but both have significant shortcomings. Although adrenal CT/MRI is widely available in various units and can effectively detect adrenal space-occupying lesions, its ability to evaluate cortical function is weak, leading to a high probability of misdiagnosis in classification diagnosis. AVS is a relatively accurate method for diagnosing aldehyde subtypes by collecting blood samples from the adrenal vein through vascular intervention to obtain information on bilateral adrenal cortical hormone secretion levels. However, as an invasive examination, AVS may lead to operational complications and pose technical challenges. In different studies and institutions, the success rate of AVS can range from 40% to 100%; due to the lack of recognized operating and evaluation standards, there are significant difficulties in the development and widespread promotion of AVS technology. Chemokine Receptor 4(CXCR4) is closely associated with the occurrence, development, and metastasis of malignant tumors, which has drawn attention in the field of radionuclide tumor imaging. Corresponding radiolabeled imaging agents have been successfully developed and utilized in clinical research. Among these, 68Ga-Pentixafor has become the most widely used CXCR4 ligand imaging agent due to its suitable half-life, high specificity, high affinity, and low background signal. Interestingly, CXCR4 is fundamentally a typical G-protein-coupled receptor (GPCR), which has been shown to be highly expressed on the cell membranes of various endocrine adenoma cells, playing a crucial role in hormone synthesis, secretion, and signal transduction. Some researchers have conducted immunohistochemical staining on adrenal adenomas and found that CXCR4 is significantly overexpressed on the cell membranes of aldosterone-producing adenoma cells, while it is either not expressed or expressed at low levels in non-functional adrenal adenomas. Based on this background, German researcher Heinze B clinically confirmed in a small sample study that 68Ga-Pentixafor Positron Emission Tomography(PET)/CT can detect aldosterone adenoma lesions in patients with primary aldosteronism. The possible mechanism is that when CXCR4 is highly expressed on the cell surface, it may respond to other regulatory factors in the body, thereby activating intracellular downstream pathways that stimulate the synthesis and secretion of aldosterone. In summary, due to its high expression in endocrine adenoma cells and its potential relationship with aldosterone synthesis and secretion, CXCR4 has become an important target in the study of primary aldosteronism. Currently, a prospective randomized comparative study of 68Ga-Pentixafor and AVS in the diagnosis of primary aldosteronism subtypes has been initiated in the Netherlands in 2022. Since 2018, I have been conducting a long-term series of studies utilizing 68Ga-Pentixafor PET/CT in patients with primary aldosteronism. Over the five years from 2018 to 2023, I have completed 68Ga-Pentixafor PET/CT imaging for more than 400 patients with primary aldosteronism, accumulating a wealth of original data and clinical experience. In the future, we plan to further explore the field of radionuclide molecular functional imaging in patients with primary aldosteronism based on our preliminary research experience and findings. Despite the significant advancements made by 68Ga-Pentixafor in the classification and diagnosis of primary aldosteronism, it is important to recognize that primary aldosteronism, as a complex systemic disease, cannot be fully elucidated solely through 68Ga-Pentixafor imaging. Furthermore, 68Ga-Pentixafor is not effective in assessing myocardial involvement in hypertensive heart disease. Beyond the organ and systemic damage caused by secondary hypertension, robust evidence indicates that aldosterone, through the activation of mineralocorticoid receptor pathways, contributes to increased vascular oxidative stress and pro-inflammatory effects, which can directly stimulate cardiac fibroblasts, leading to the development of myocardial fibrosis and hypertrophy. This significantly elevates the risk of cardiovascular events in patients and is one of the leading causes of mortality in individuals with primary aldosteronism. A cross-sectional study involving 2,612 hypertensive patients in China observed a notable increase in the risk of cardiovascular disease associated with primary aldosteronism compared to hypertensive patients with normal aldosterone levels (odds ratio of 2.57). In another study comparing patients with primary aldosteronism to matched hypertensive controls, it was found that the incidence of stroke was four times higher, the risk of myocardial infarction was increased by 6.5 times, and the prevalence of atrial fibrillation was twelve times greater in patients with primary aldosteronism. Research indicates that early intervention can significantly reduce the incidence of cardiovascular events in these patients. Therefore, in addition to classification and diagnosis, early and comprehensive assessment of the extent of cardiovascular and other organ damage in patients with primary aldosteronism holds substantial clinical significance. Myocardial fibrosis is a common pathological change that occurs in the progression of most cardiovascular diseases, often manifesting early and persisting throughout the disease course. It primarily results from the excessive proliferation of cardiac fibroblasts and their transformation into myofibroblasts, leading to significant extracellular matrix deposition in the myocardial interstitium, which subsequently causes cardiac remodeling. Myocardial fibrosis is frequently associated with impaired cardiac contractile and diastolic function, arrhythmias, and adverse cardiovascular events. The probability of asymptomatic myocardial fibrosis in patients with primary aldosteronism can reach up to 70% in the early stages of the disease. Fibrosis assessment is a crucial imaging target for providing cardiac risk stratification in these patients. Research has shown that the increased level of myocardial fibrosis in patients with primary aldosteronism may be reversible through adrenalectomy, significantly reducing the incidence of cardiovascular events. While pharmacological treatment can also partially reverse myocardial hypertrophy and fibrosis, the cardiovascular outcomes are generally not as favorable as those in patients who undergo surgical treatment. One possible reason for this discrepancy is that the selection of medication dosages has not incorporated effective assessment indicators for the degree of cardiovascular damage, leading to insufficient antagonistic effects of the medication against the cardiovascular toxicity of aldosterone. In addition to lowering blood pressure, treatment targeting excess aldosterone is equally important for patients with primary aldosteronism. Due to the current lack of specific therapeutic methods for myocardial fibrosis, early exploration and intervention during the active phase of fibroblast activity and the reversible stage of fibrosis become increasingly important. Early investigation and intervention in the level of myocardial fibrosis in patients with primary aldosteronism can partially reverse fibrosis levels, which is significant for effectively identifying and controlling myocardial fibrosis in the prevention and treatment of cardiac diseases, as well as improving the quality of life for these patients. Endomyocardial biopsy and fibrosis staining are considered the gold standard for diagnosing myocardial fibrosis. By analyzing and quantifying the interstitial collagen in biopsy samples, one can estimate the extent of myocardial fibrosis. However, this invasive procedure carries significant risks, is technically challenging, and poses difficulties in accurately targeting affected myocardial tissue, making it unsuitable for widespread clinical application. A range of established diagnostic techniques allows for non-invasive assessment of myocardial fibrosis, including serum biomarker tests, echocardiography, and cardiac magnetic resonance (CMR) imaging. In terms of biochemical blood tests, several serum biomarkers that reflect fibrotic activity are available, but they lack cardiac specificity and may also be elevated in cases of fibrosis in other parts of the body. Echocardiography, as a non-invasive and straightforward examination, has become an important tool for detecting cardiac diseases; however, it cannot accurately display pathological changes within the myocardium and is typically used for supplementary evaluation of myocardial fibrosis. CMR can assess the anatomical and functional status of the heart, particularly through late gadolinium enhancement (LGE) and functional CMR techniques, which include native T1 mapping and extracellular volume (ECV) measurements, allowing for localization and quantification of fibrotic lesions. Nevertheless, there are limitations to CMR. Firstly, it can only identify myocardium that has already undergone fibrosis and is less effective at recognizing the interstitial changes in actively fibrosing myocardium, thus failing to detect the ongoing remodeling process. Secondly, since it requires a reference of normal myocardium, it has limitations in detecting diffuse myocardial fibrosis. Additionally, the results may not be entirely specific to fibrosis, as they can overlap with manifestations of myocardial edema, inflammation, and amyloid deposition. Furthermore, gadolinium-based contrast agents carry risks of renal impairment and allergic reactions. The specific expression of fibroblast activation protein (FAP) on activated fibroblasts has garnered significant attention in recent years. In 2018, the Haberkorn team from Heidelberg University in Germany published an important study in the Journal of Nuclear Medicine regarding radiolabeled targeted FAP-specific enzyme inhibitors (FAPI) for molecular imaging. These radiolabeled compounds exhibit favorable pharmacokinetic properties and high affinity for FAP, demonstrating great potential in the early imaging studies of tumor-associated fibroblasts. Their research indicated that 68Ga-FAPI shows extremely high detection sensitivity in various epithelial-derived tumor lesions. Given that inflammation-related fibroblasts can be observed with high FAP expression while normal myocardial tissue exhibits almost no FAP expression, 68Ga-FAPIs are currently being utilized in clinical studies for various cardiovascular diseases, including acute myocardial infarction, hypertrophic cardiomyopathy, dilated cardiomyopathy, and heart failure. They are considered biomarkers for myocardial injury, fibrotic activity, and matrix remodeling. This characteristic of FAP may provide a robust target for the early diagnosis and assessment of myocardial fibrosis in patients with primary aldosteronism. This approach may allow for highly specific imaging of fibrotic activity for the first time, providing a basis for early fibrosis detection and distinguishing between active disease and end-stage disease. The novel molecular receptor imaging method for fibrosis, utilizing FAPI tracers, opens new avenues for a deeper understanding of tissue fibrosis. In recent years, the advent of simultaneous PET/MR technology has marked a significant breakthrough in the field of imaging. PET/MR is an advanced integration of PET and MR, allowing for both PET and MR examinations to be completed in a single scan. By combining the ultra-high-resolution images from MR with the cellular metabolic and molecular changes captured by PET, this technology offers a new imaging paradigm that achieves a synergistic effect greater than the sum of its parts. Building on this foundation, the combination of simultaneous PET and CMR represents the latest advancement in non-invasive diagnostics for cardiac diseases. This approach enables the simultaneous acquisition of detailed anatomical structures of the heart, myocardial perfusion levels, cardiac function assessment, delayed enhancement information, functional MRI data, and PET metabolic parameters, providing greater advantages compared to separate PET and CMR systems. The use of 68Ga-FAPI PET/CMR has the potential to integrate structural and functional parameters, emerging as a new standard for detecting early myocardial fibrosis and cardiovascular risk stratification in patients with primary aldosteronism, ultimately serving as a direct endpoint for evaluating treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Research Group Inclusion Criteria - (1) Patients must be over 18 years of age. (2) Patients diagnosed by an endocrinologist as highly suspected or confirmed cases of primary aldosteronism according to the guidelines of the Endocrine Society will be included.

1. The criteria for high suspicion are as follows:

   ① Persistent hypertension >160/100 mmHg, especially resistant hypertension (blood pressure remains >140/90 mmHg despite treatment with three or more antihypertensive medications) accompanied by hypokalemia (serum potassium concentration <3.5 mmol/L); or ② Drug-resistant hypokalemia with or without hypertension; or ③ Persistent hypertension with plasma aldosterone concentration (PAC) >15 ng/dl and a plasma aldosterone-renin ratio (ARR) ≥30 (ng/dl)/(ng/ml/h) (when plasma renin activity <0.1 ng/ml/h, it is calculated as 0.1 ng/ml/h).
2. The criteria for confirming primary aldosteronism are as follows:

Under the conditions of high suspicion, a positive result from the captopril challenge test (CCT) must be met. The principles, examination process, and methods for positive assessment of the CCT are as follows:

* Principle: Captopril is an angiotensin-converting enzyme inhibitor that can suppress the renin-angiotensin-aldosterone system in normal individuals, thereby reducing aldosterone secretion. However, it has no significant inhibitory effect on patients with autonomous aldosterone secretion, such as those with primary aldosteronism.

  * Examination method: Discontinue aldosterone antagonists and angiotensin-converting enzyme inhibitors for 1-2 weeks. On the day of the test, the patient should remain seated or supine for at least 4 hours, then orally administer 25 mg of captopril, and maintain the same position for 2 hours before drawing blood to measure PAC and PRA levels.

    * Evaluation of test results: Calculate the change rate of PAC before and after the test, as well as the ARR value after the test. Based on published data, a reduction in PAC of <30% compared to pre-test levels or an ARR value >46.2 after the CCT is considered a diagnostic threshold for a positive test result.

      (3) Imaging studies indicate the presence of unilateral or bilateral adrenal nodules or nodular hyperplasia in the patient.

      (4) Prior to enrollment, patients will undergo echocardiography, and the results will be recorded. If left ventricular hypertrophy is indicated, the patient will be included in the primary aldosteronism group with myocardial hypertrophy; otherwise, they will be included in the primary aldosteronism group without myocardial hypertrophy. Control Group Inclusion Criteria (1) The patient is over 18 years of age.

      (2) The systolic blood pressure is greater than or equal to 140 mmHg or the diastolic blood pressure is greater than or equal to 90 mmHg.

      (3) The patient's biochemical tests indicate normal adrenal hormone secretion. (4) There are no identifiable causes of secondary hypertension. (5) Imaging studies suggest the presence of unilateral or bilateral adrenal nodules or nodular hyperplasia in the patient.

      (6) the patient undergoes a cardiac ultrasound before enrollment, and the results are recorded. If the ultrasound indicates left ventricular hypertrophy, the patient is included in the primary hypertension group with myocardial hypertrophy; otherwise, they are included in the primary hypertension group without myocardial hypertrophy.

Exclusion Criteria:

(1) Children, pregnant and lactating women, etc; (2) Patients with poor autonomous behavioral ability (such as inability to lie flat), severe claustrophobia, and critically ill patients requiring life support who are unable to cooperate in completing the examination; (3) Patients with severe liver and kidney failure; (4) Patients with a history of myocardial infarction, cardiomyopathy, myocarditis, or congenital heart disease in the past; (5) Patients who can not successfully undergo CMR examination, such as arrhythmia or inability to hold their breath. (6) Patients with other conditions that are not suitable for this examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion and exclusion criteria and are willing to follow the research process.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
positive lesion of adrenal gland | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  The first step is to visually evaluate the image by comparing the tracer uptake of adrenal lesions with adjacent and contralateral adrenal tissues. The evaluation results are as follows: ① PET-positive lesions: Adrenal lesions with significantly higher levels of radioactive uptake than normal adrenal tissue; ② PET-negative lesions: Adrenal lesions with similar or lower levels of radioactive uptake compared to normal adrenal tissue. If the bilateral adrenal glands show multiple nodular thickening without obvious normal adrenal tissue, the radiation level in the non-nodular thickening area can be used as a reference. If there are focal adrenal nodules with increased radioactive uptake, it is still considered a positive lesion.
Calculate standardized uptake value on 68Ga-Pentixafor PET | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  In PET/MR imaging, the first step is to identify the adrenal lesion area based on morphological characteristics. Using the reconstruction software from United Imaging, I delineate the region of interest (ROI) within the adrenal lesion area. Additionally, I outline the ROI for normal liver tissue and other normal tissues in the body. The liver ROI is defined as a sphere with a diameter of 2 centimeters, typically selected from the liver tissue at the same level as the right adrenal gland. The ROI for normal adrenal tissue is a sphere with a diameter of 0.6 to 0.8 centimeters, with the contralateral normal adrenal tissue being the primary choice, followed by the ipsilateral normal adrenal tissue. Non-nodular areas of adrenal thickening are only considered when no normal adrenal tissue is available. Subsequently, the software automatically generates the maximum standardized uptake value (SUVmax) for the adrenal lesion, the mean standardized uptake value (SUVmean) for normal liver tissue.
Left ventricular ejection fraction（LVEF） | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Analyzing LVEF on CMR images.
systolic wall thickening(Δ T%) | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Analyzing the thickening rate of the ventricular wall in each segment of the myocardium.
Calculate maximum standardized uptake value of the heart on 68Ga-FAPI-04 PET | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Use the American Heart Association's 17 segment method to evaluate for increased radioactive uptake in each segment of myocardium, record the number of positive uptake segments, then delineate the ROI value and calculate SUVmax.

IPD SHARING:
Plan to Share IPD: No
For the protection of patient privacy, we will not share patient information, but other researchers can apply through the project contact person if they have reasonable reasons.